CLINICAL TRIAL: NCT00968578
Title: Effects of Pre-operative Methylprednisolone (125mg iv) After Total Knee Arthroplasty: A Prospective, Randomized, Double-blind, Placebo-controlled Trail
Brief Title: Effects of Methylprednisolone After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-C-2008-134; 2009-41-3786
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Sleeping Quality; Fatigue; Inflammatory Response
Keywords: Knee arthroplasty; Methylprednisolone; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Fatigue | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylprednisolone (Active Comparator): Methylprednisolone 125 mg iv pre-operatively
  Interventions: Drug: Methylprednisolone
- Saline (Placebo Comparator): Saline iv pre-operatively in equivalent volume (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone 125 mg iv pre-operatively
  Arms: Methylprednisolone
Drug: Placebo — Saline iv pre-operatively in equivalent volume (placebo)
  Arms: Saline

SUMMARY:
The purpose of the study is to compare the effects of pre-operative methylprednisolone (125mg iv) versus placebo on postoperative outcome after knee arthroplasty.

The hypothesis is that pre-operative methylprednisolone (125mg iv) will reduce pain and improve outcome.

DETAILED DESCRIPTION:
In spite of being one of the last century's most successful surgical procedures in treatment of advanced osteoarthritis total knee arthroplasty is still associated with postoperative pain and delayed rehabilitation. We therefore decided to evaluate the effects of pre-operative methylprednisolone (125mg iv) versus placebo on postoperative outcome in a well defined fast-track setup after knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Elective total knee arthroplasty
* Able to speak and understand danish
* Able to give informed consent

Exclusion Criteria:

* Alcohol or medical abuse
* Allergies to local anesthetics or methylprednisolone
* Age < 18 years
* Daily use of opioids or glucocorticoids
* Pregnancy or breastfeeding (fertile women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours + follow up

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 48 hours + follow up
Sleeping quality | 48 hours + follow up
Inflammatory response | 48 hours + follow up
Additional analgetics, antinausea agents and sleeping medicine | 48 hours + follow up
Time in hospital | Until discharge
Fatigue | 48 hours + follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Lunn TH, Kristensen BB, Andersen LO, Husted H, Otte KS, Gaarn-Larsen L, Kehlet H. Effect of high-dose preoperative methylprednisolone on pain and recovery after total knee arthroplasty: a randomized, placebo-controlled trial. Br J Anaesth. 2011 Feb;106(2):230-8. doi: 10.1093/bja/aeq333. Epub 2010 Dec 3. PMID 21131371